CLINICAL TRIAL: NCT04627116
Title: A Multiple-Dose, Safety and Tolerability、PK/PD Study of Tecarfarin in Healthy Chinese Volunteers
Brief Title: An Ascending, Multiple-Dose, Safety and Tolerability Study of Tecarfarin in Healthy Chinese Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ZK-TEK-201905
Record Dates: First submitted 2020-09-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Healthy Chinese Volunteers
MeSH Terms: interventions — tecarfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tecarfarin 10mg (Experimental)
  Interventions: Drug: Tecarfarin
- Tecarfarin 20mg (Experimental)
  Interventions: Drug: Tecarfarin
- Tecarfarin 30mg (Experimental)
  Interventions: Drug: Tecarfarin
- Tecarfarin 40mg (Experimental)
  Interventions: Drug: Tecarfarin

INTERVENTIONS:
Drug: Tecarfarin — Ten (10) healthy Chinese subjects received once-daily doses of Tecarfarin on fasting every morning for 14 days.

SUMMARY:
The subjects will be admitted to the Phase I Clinical Research Center on day -1. Subjects received once-daily doses of Tecarfarin for up to 14 days.Subjects can leave the Phase I Clinical Research Center on the day 21.And returned to the research center for follow-up on the day 28 and 35.

ELIGIBILITY:
Inclusion Criteria:

1) the subjects were fully aware of the purpose, nature, methods and possible adverse reactions of the trial, voluntarily act as subjects, and sign an informed consent form before the commencement of any research process.

2）Healthy volunteers between the ages of 18 to 50 years old (inclusive). 3）Weight: male ≥ 50.0kg, female ≥ 45.0kg; Body Mass Index (BMI) ≥19 and ≤ 24 kg/m2.

4) The physical examination, vital sign measurements, clinical laboratory assessments hematology, clinical chemistry, or urinalysis, etc.) and 12-lead ECG were judged normal, or abnormal without clinical significance by the investigators.

Exclusion Criteria:

1. Positive test results for HIV, syphilis antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV Ab) at Screening.

2) Dysphagia or documented history of any gastrointestinal disorders that affect drug absorption.

3) Subjects with difficulty in venipuncture, those who cannot tolerate venipuncture, and those who have a history of needlesickness and bloodsickness.

4) Positive tests for urine drugs of abuse at Screening or a history of drug or alcohol abuse/dependence.

5) Use of tobacco products 3 months before screening. 6）Heavy tea, coffee and / or caffeinated drinks (more than 8 cups, 1 cup = 250 mL) drinker per day within 3 months prior to screening.

7）Subjects who drunk frequently within 6 months prior to screening (intake of more than 14 units of alcohol per week. A unit is 360 mL beer, 45 mL of 40% liquor or 150 mL wine).

8）Any out-of-normal-range PT, aPTT, TT, FIB,INR, protein C, protein S or coagulation factors II, VII, X at screening.

9）History of cardiovascular, renal, pulmonary, nervous system, liver and/or endocrine disease.

10）Documented history of bleeding diathesis, coagulopathy, or inherited disorders of coagulation.

11）Evidence of active bleeding, including but not limited to gastrointestinal bleeding (hematemesis, hematochezia, positive fecal occult blood), urinary tract bleeding, mucosal bleeding (gingival, epistaxis) and unexplained subcutaneous bleeding or ecchymosis.

12）Participation in a previous clinical trial within 3 months prior to Screening.

13）Clinically significant surgical procedure within 4 weeks prior to Screening or planned to undergo surgery during the study period.

14) Clinically significant blood loss or blood donation > 550 ml within 3 months prior to Screening.

15）Taking any medication 14 days prior to Screening. 16）Known allergy or hypersensitivity to warfarin or the investigational product.

17）Pregnancy or Lactation. 18）Female subjects cannot avoid menstruation during administration. 19）subjects of childbearing age are not guaranteed to have no fertility plan, sperm donation, egg donation plan and voluntary use of non-drug contraceptive measures (including subcutaneous injection of contraceptive, contraceptive injections, subcutaneous implantation of contraceptives, local contraceptives such as spermicide, etc.) from two weeks before screening to 6 months after the end of the trial.

20）Investigator would make the subject unsuitable for the study or put them at additional risks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study was to evaluate the safety and tolerability of Tecarfarin when administered as rising multiple oral doses to healthy Chinese volunteers. | doses of Tecarfarin for up to 14 days.
  Subjects received once-daily doses of Tecarfarin for up to 14 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou Q, Wang Z, Wang H, Chen Z, Li X, Dai X, Zhang Y, Yu X, Zhou R, Hu W. Safety and Tolerability of Tecarfarin (ATI-5923) in Healthy Chinese Volunteers: Multiple Oral Dose-Escalation Phase I Trial. Am J Cardiovasc Drugs. 2023 Jan;23(1):101-112. doi: 10.1007/s40256-022-00562-5. Epub 2023 Jan 9. PMID 36622539